CLINICAL TRIAL: NCT03612986
Title: Double Blind, Placebo Controlled Trial to Evaluate the Effects of a Nutraceutical Containing High-Molecular-Weight Hyaluronic Acid (HA) and Acetyl-11-Keto-Beta-Boswellic Acid (AKBA) in Patients Affected by Knee Osteoarthritis
Brief Title: Clinical Trial to Evaluate the Effects of a Nutraceutical in Patients Affected by Knee Osteoarthritis
Acronym: SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: River Pharma S.r.l. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPRPH/0118/FS
Record Dates: First submitted 2018-07-04; First posted 2018-08-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Active comparator SYALOX® 300 Plus (Active Comparator): Active Nutraceutical containing HA and AKBA (SYALOX® 300 Plus)
  1 tablet/day, oral administration
  Interventions: Dietary Supplement: SYALOX® 300 Plus
- B: Placebo (Placebo Comparator): Placebo
  1 tablet/day, oral administration
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: SYALOX® 300 Plus — Reduction of pain and improvement of the knee mobility in patients affected by knee osteoarthritis
  Arms: A: Active comparator SYALOX® 300 Plus
Dietary Supplement: Placebo — Placebo comparator. No chemical effect expected
  Arms: B: Placebo

SUMMARY:
Double blind, placebo controlled trial to evaluate the effects of a nutraceutical containing high-molecular-weight hyaluronic acid (HA) and acetyl-11-keto-beta-boswellicacid (AKBA) in patients affected by knee osteoarthritis.

DETAILED DESCRIPTION:
The primary objective of the trial is to assess the feasibility of implementing Ultrasonography and Range of Motion (ROM) as objective measurements to correlate the improvement of the knee mobility with the pain reduction of the affected knee in the patients assuming nutraceutical containing hyaluronic acid (HA).

The secondary objectives of the trial are:

* to assess the feasibility of implementing Actigraphy as objective measurements to correlate the improvement of the knee mobility with the pain reduction (optional).
* to evaluate the enrollment rate in one month.

The explorative objectives of the trial are:

• Preliminary data on efficacy of the tested product.

ELIGIBILITY:
Inclusion Criteria:

* Any gender and age from 45 to 70 years
* Symptomatic osteoarthritis (OA) of the knee with mild joint discomfort for at least 6 months prior to enrollment, following ACR criteria with history and physical examination(44). Subjects diagnosed with bilateral knee OA will be asked to specify the most affected knee at baseline, and this knee will be evaluated throughout the study period.
* Available confirmatory X-ray (performed within the previous 6 months) diagnosis (Kellgren/Lawrence score 2) at the evaluated knee joint(45).
* Subjects experienced pain for at least 15 of the 30 days prior to the start of the study.

Exclusion Criteria:

* Subjects who have any inflammatory arthritic condition (different from the OA of the knee), fibromyalgia, multiple sclerosis or autoimmune disorder.
* Treatment with oral corticosteroids within 4 weeks before screening.
* Intra-articular injections of HA or corticosteroids in the target joint within 3 months before screening.
* Treatment with anti-inflammatory or chondroprotective drugs (chondroitin sulfate, glucosamine, methylsulfonylmethane, HA, diacerein) 2 weeks before the selection.
* HA-containing nutritional supplements or cosmetics during the month before the study.
* Previous surgical treatment of knee joint(s) or its necessity necessity for osteoarthritis (high tibial osteotomy, arthroplasty); complication(s) necessary for hospitalization and surgical treatment.
* Significant injury to the target joint within the past 6 months prior to screening (identified from medical history).
* Subjects following an energy-restricted diet for weight loss.
* Pregnant women, nursing mothers, or women (only if childbearing potential) not using adequate methods of contraception.
* Subjects with cardiovascular, hepatic, renal, respiratory, or hematologic illness, or other medical or psychiatric condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the course of the study.
* Participation in an interventional clinical study in the previous 30 days.
* Presence of any clinically significant medical condition judged by the investigator to preclude the patient's inclusion in the study.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) results at rest. Change is being assessed. | week 0, 4 and 16
  Change in Visual Analogue Scale (VAS) results at rest, measured in mm
Knee Range of Motion (ROM) results measured by goniometer. Change is being assessed. | week 0, 4 and 16
  Change in Range of Motion (ROM) results, measured in grades by goniometer.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) results at moving. Change is being assessed. | week 0, 4 and 16
  Change in Visual Analogue Scale (VAS) results at moving, measured in mm
Visual Analogue Scale (VAS) results on pressing. Change is being assessed. | week 0, 4 and 16
  Change in Visual Analogue Scale (VAS) results at pressing, measured in mm
Ultrasonography parameters results. Change is being assessed. | week 0 and 16
  Change of presence or absence of Synovial fluid, Articular cartilage damage, Medial meniscal protrusion, Lateral meniscal protrusion, Medial osteophytes, Lateral osteophytes, Enthesopathies, Effusion is being assessed.
Knee injury and Osteoarthritis Outcome Score (KOOS). Change is being assessed. | week 0, 4 and 16
  Change in parameters of quality of life will be assessed through Knee injury and Osteoarthritis Outcome Score (KOOS).
Index of Severity for Osteoarthritis of the Knee by Lequesne et al. Change is being assessed. | week 0, 4 and 16
  Change in parameters of quality of life will be assessed through Index of Severity for Osteoarthritis of the Knee by Lequesne et al.
Knee movement results using an actimeter (accelerometer). Change is being assessed. | week 0 and 16
  Knee movement based on acceleration results using an actimeter, device based on an accelerometer. The results will be measured in meter/second squared (m/s2) Change is being assessed.

OTHER OUTCOMES:
Safety outcomes assessed by number of adverse events (AE)/serious adverse events (SAE) | day 0, week 4 and 16
  Adverse events (AE)/serious adverse events (SAE) (number of events occured, related to the investigational product administration)
Safety assessment based on rescue medication (Paracetamol 500mg) administration | day 0, week 4 and 16
  Safety assessed by the number of rescue medication tablets administered daily.

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Andor, MD, Principal Investigator — MEDICALI'S
Locations (1):
- Opera Contract Research Organization S.r.l., Timișoara, Timiș County, Romania

REFERENCES:
- [Background] Bhatia D, Bejarano T, Novo M. Current interventions in the management of knee osteoarthritis. J Pharm Bioallied Sci. 2013 Jan;5(1):30-8. doi: 10.4103/0975-7406.106561. PMID 23559821
- [Background] Carvalho NA, Bittar ST, Pinto FR, Ferreira M, Sitta RR. Manual for guided home exercises for osteoarthritis of the knee. Clinics (Sao Paulo). 2010 Jun;65(8):775-80. doi: 10.1590/s1807-59322010000800006. PMID 20835554
- [Background] Voelker R. Few adults with knee osteoarthritis meet national guidelines for physical activity. JAMA. 2011 Oct 5;306(13):1428, 1430. doi: 10.1001/jama.2011.1388. No abstract available. PMID 21972300
- [Background] Pai YC, Chang HJ, Chang RW, Sinacore JM, Lewis JL. Alteration in multijoint dynamics in patients with bilateral knee osteoarthritis. Arthritis Rheum. 1994 Sep;37(9):1297-304. doi: 10.1002/art.1780370905. PMID 7945492
- [Background] Cutolo M, Berenbaum F, Hochberg M, Punzi L, Reginster JY. Commentary on recent therapeutic guidelines for osteoarthritis. Semin Arthritis Rheum. 2015 Jun;44(6):611-7. doi: 10.1016/j.semarthrit.2014.12.003. Epub 2014 Dec 24. PMID 25677861
- [Background] Bruyere O, Cooper C, Pelletier JP, Maheu E, Rannou F, Branco J, Luisa Brandi M, Kanis JA, Altman RD, Hochberg MC, Martel-Pelletier J, Reginster JY. A consensus statement on the European Society for Clinical and Economic Aspects of Osteoporosis and Osteoarthritis (ESCEO) algorithm for the management of knee osteoarthritis-From evidence-based medicine to the real-life setting. Semin Arthritis Rheum. 2016 Feb;45(4 Suppl):S3-11. doi: 10.1016/j.semarthrit.2015.11.010. Epub 2015 Dec 2. PMID 26806188
- [Background] Bruyere O, Burlet N, Delmas PD, Rizzoli R, Cooper C, Reginster JY. Evaluation of symptomatic slow-acting drugs in osteoarthritis using the GRADE system. BMC Musculoskelet Disord. 2008 Dec 16;9:165. doi: 10.1186/1471-2474-9-165. PMID 19087296
- [Background] Bannuru RR, Schmid CH, Kent DM, Vaysbrot EE, Wong JB, McAlindon TE. Comparative effectiveness of pharmacologic interventions for knee osteoarthritis: a systematic review and network meta-analysis. Ann Intern Med. 2015 Jan 6;162(1):46-54. doi: 10.7326/M14-1231. PMID 25560713
- [Background] Navarro-Sarabia F, Coronel P, Collantes E, Navarro FJ, de la Serna AR, Naranjo A, Gimeno M, Herrero-Beaumont G; AMELIA study group. A 40-month multicentre, randomised placebo-controlled study to assess the efficacy and carry-over effect of repeated intra-articular injections of hyaluronic acid in knee osteoarthritis: the AMELIA project. Ann Rheum Dis. 2011 Nov;70(11):1957-62. doi: 10.1136/ard.2011.152017. Epub 2011 Aug 17. PMID 21852252
- [Background] Waddell DD, Bricker DC. Total knee replacement delayed with Hylan G-F 20 use in patients with grade IV osteoarthritis. J Manag Care Pharm. 2007 Mar;13(2):113-121. doi: 10.18553/jmcp.2007.13.2.113. PMID 17330972
- [Background] Reed RK, Townsley MI, Laurent TC, Taylor AE. Hyaluronan flux from cat intestine: changes with lymph flow. Am J Physiol. 1992 Feb;262(2 Pt 2):H457-62. doi: 10.1152/ajpheart.1992.262.2.H457. PMID 1539704
- [Background] Balogh L, Polyak A, Mathe D, Kiraly R, Thuroczy J, Terez M, Janoki G, Ting Y, Bucci LR, Schauss AG. Absorption, uptake and tissue affinity of high-molecular-weight hyaluronan after oral administration in rats and dogs. J Agric Food Chem. 2008 Nov 26;56(22):10582-93. doi: 10.1021/jf8017029. PMID 18959406
- [Background] Hisada N, Satsu H, Mori A, Totsuka M, Kamei J, Nozawa T, Shimizu M. Low-molecular-weight hyaluronan permeates through human intestinal Caco-2 cell monolayers via the paracellular pathway. Biosci Biotechnol Biochem. 2008 Apr;72(4):1111-4. doi: 10.1271/bbb.70748. Epub 2008 Apr 7. PMID 18391466
- [Background] Laznicek M, Laznickova A, Cozikova D, Velebny V. Preclinical pharmacokinetics of radiolabelled hyaluronan. Pharmacol Rep. 2012;64(2):428-37. doi: 10.1016/s1734-1140(12)70784-3. PMID 22661195
- [Background] Altman RD, Manjoo A, Fierlinger A, Niazi F, Nicholls M. The mechanism of action for hyaluronic acid treatment in the osteoarthritic knee: a systematic review. BMC Musculoskelet Disord. 2015 Oct 26;16:321. doi: 10.1186/s12891-015-0775-z. PMID 26503103
- [Background] du Souich P. Absorption, distribution and mechanism of action of SYSADOAS. Pharmacol Ther. 2014 Jun;142(3):362-74. doi: 10.1016/j.pharmthera.2014.01.002. Epub 2014 Jan 21. PMID 24457028
- [Background] Oe M, Tashiro T, Yoshida H, Nishiyama H, Masuda Y, Maruyama K, Koikeda T, Maruya R, Fukui N. Oral hyaluronan relieves knee pain: a review. Nutr J. 2016 Jan 27;15:11. doi: 10.1186/s12937-016-0128-2. PMID 26818459
- [Background] Yasui T, Akatsuka M, Tobetto K, Hayaishi M, Ando T. The effect of hyaluronan on interleukin-1 alpha-induced prostaglandin E2 production in human osteoarthritic synovial cells. Agents Actions. 1992 Sep;37(1-2):155-6. doi: 10.1007/BF01987905. PMID 1456177
- [Background] Homandberg GA, Ummadi V, Kang H. The role of insulin-like growth factor-I in hyaluronan mediated repair of cultured cartilage explants. Inflamm Res. 2004 Aug;53(8):396-404. doi: 10.1007/s00011-004-1276-y. Epub 2004 Aug 10. PMID 15316671
- [Background] Wang CT, Lin YT, Chiang BL, Lin YH, Hou SM. High molecular weight hyaluronic acid down-regulates the gene expression of osteoarthritis-associated cytokines and enzymes in fibroblast-like synoviocytes from patients with early osteoarthritis. Osteoarthritis Cartilage. 2006 Dec;14(12):1237-47. doi: 10.1016/j.joca.2006.05.009. Epub 2006 Jun 30. PMID 16806998
- [Background] Waller KA, Zhang LX, Fleming BC, Jay GD. Preventing friction-induced chondrocyte apoptosis: comparison of human synovial fluid and hylan G-F 20. J Rheumatol. 2012 Jul;39(7):1473-80. doi: 10.3899/jrheum.111427. Epub 2012 Jun 1. PMID 22660808
- [Background] Bernad Pineda M. Current status of symptomatic slow-acting drugs for osteoarthritis (SYSADOAs) in Spain. Reumatol Clin. 2016 Jul-Aug;12(4):181-3. doi: 10.1016/j.reuma.2016.03.012. Epub 2016 Apr 18. No abstract available. English, Spanish. PMID 27101743
- [Background] Tashiro T, Seino S, Sato T, Matsuoka R, Masuda Y, Fukui N. Oral administration of polymer hyaluronic acid alleviates symptoms of knee osteoarthritis: a double-blind, placebo-controlled study over a 12-month period. ScientificWorldJournal. 2012;2012:167928. doi: 10.1100/2012/167928. Epub 2012 Nov 20. PMID 23226979
- [Background] Nagaoka I, Nabeshima K, Murakami S, Yamamoto T, Watanabe K, Tomonaga A, Yamaguchi H. Evaluation of the effects of a supplementary diet containing chicken comb extract on symptoms and cartilage metabolism in patients with knee osteoarthritis. Exp Ther Med. 2010 Sep;1(5):817-827. doi: 10.3892/etm.2010.114. Epub 2010 Jul 12. PMID 22993606
- [Background] Sanchez J, Bonet ML, Keijer J, van Schothorst EM, Molller I, Chetrit C, Martinez-Puig D, Palou A. Blood cells transcriptomics as source of potential biomarkers of articular health improvement: effects of oral intake of a rooster combs extract rich in hyaluronic acid. Genes Nutr. 2014 Sep;9(5):417. doi: 10.1007/s12263-014-0417-3. Epub 2014 Jul 15. PMID 25024048
- [Background] D'Agostino MA, Conaghan P, Le Bars M, Baron G, Grassi W, Martin-Mola E, Wakefield R, Brasseur JL, So A, Backhaus M, Malaise M, Burmester G, Schmidely N, Ravaud P, Dougados M, Emery P. EULAR report on the use of ultrasonography in painful knee osteoarthritis. Part 1: prevalence of inflammation in osteoarthritis. Ann Rheum Dis. 2005 Dec;64(12):1703-9. doi: 10.1136/ard.2005.037994. Epub 2005 May 5. PMID 15878903
- [Background] Hartung W, Kellner H, Strunk J, Sattler H, Schmidt WA, Ehrenstein B, Fleck M, Backhaus M. Development and evaluation of a novel ultrasound score for large joints in rheumatoid arthritis: one year of experience in daily clinical practice. Arthritis Care Res (Hoboken). 2012 May;64(5):675-82. doi: 10.1002/acr.21574. PMID 22183834
- [Background] Serban O, Porojan M, Deac M, Cozma F, Solomon C, Lenghel M, Micu M, Fodor D. Pain in bilateral knee osteoarthritis - correlations between clinical examination, radiological, and ultrasonographical findings. Med Ultrason. 2016 Sep;18(3):318-25. doi: 10.11152/mu.2013.2066.183.pin. PMID 27622408
- [Background] Wu PT, Shao CJ, Wu KC, Wu TT, Chern TC, Kuo LC, Jou IM. Pain in patients with equal radiographic grades of osteoarthritis in both knees: the value of gray scale ultrasound. Osteoarthritis Cartilage. 2012 Dec;20(12):1507-13. doi: 10.1016/j.joca.2012.08.021. Epub 2012 Sep 1. PMID 22944523
- [Background] Yoshimura M, Aoba Y, Watari T, Momomura R, Watanabe K, Tomonaga A, Matsunaga M, Suda Y, Lee WY, Asai K, Yoshimura K, Nakagawa T, Yamamoto T, Yamaguchi H, Nagaoka I. Evaluation of the effect of a chicken comb extract-containing supplement on cartilage and bone metabolism in athletes. Exp Ther Med. 2012 Oct;4(4):577-580. doi: 10.3892/etm.2012.646. Epub 2012 Jul 24. PMID 23170108
- [Background] Yoshimura M, Aoba Y, Naito K, Watari T, Murakami S, Yoshimura K, Nakagawa T, Yamamoto T, Yamaguchi H, Nagaoka I. Effect of a chicken comb extract-containing supplement on subclinical joint pain in collegiate soccer players. Exp Ther Med. 2012 Mar;3(3):457-462. doi: 10.3892/etm.2011.431. Epub 2011 Dec 23. PMID 22969911
- [Background] Steins D, Dawes H, Esser P, Collett J. Wearable accelerometry-based technology capable of assessing functional activities in neurological populations in community settings: a systematic review. J Neuroeng Rehabil. 2014 Mar 13;11:36. doi: 10.1186/1743-0003-11-36. PMID 24625308
- [Background] Yang CC, Hsu YL. A review of accelerometry-based wearable motion detectors for physical activity monitoring. Sensors (Basel). 2010;10(8):7772-88. doi: 10.3390/s100807772. Epub 2010 Aug 20. PMID 22163626
- [Background] Trudeau J, Van Inwegen R, Eaton T, Bhat G, Paillard F, Ng D, Tan K, Katz NP. Assessment of pain and activity using an electronic pain diary and actigraphy device in a randomized, placebo-controlled crossover trial of celecoxib in osteoarthritis of the knee. Pain Pract. 2015 Mar;15(3):247-55. doi: 10.1111/papr.12167. Epub 2014 Feb 5. PMID 24494935
- [Background] Wylde V, Lenguerrand E, Brunton L, Dieppe P, Gooberman-Hill R, Mann C, Blom AW. Does measuring the range of motion of the hip and knee add to the assessment of disability in people undergoing joint replacement? Orthop Traumatol Surg Res. 2014 Apr;100(2):183-6. doi: 10.1016/j.otsr.2013.09.016. Epub 2014 Feb 17. PMID 24556210
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- See also: Proverb resources: Ashanti Proverbs from Ghana — http://cogweb.ucla.edu/Discourse/Proverbs/Ashanti.html